CLINICAL TRIAL: NCT06010056
Title: PCA Ketamine-Morphine Versus PCA Morphine as Post-Operative Analgesia in Colorectal Surgery.
Brief Title: PCA Ketamine-Morphine VS PCA Morphine as Post-Operative Analgesia in Colorectal Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JEP-2018-092
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Ketamine; Morphine
Keywords: Colorectal surgery; patient-controlled analgesia; postoperative pain management
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Intervention Model Description: Participants were randomly allocated into either Group A or Group B by computer-generated randomization a day before planned surgery.
  Group A will receive PCA ketamine-morphine 0.5 mg/ml in 1:1 ratio while group B will receive PCA morphine 1mg/ml.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patients, nurses who cared for the patients, the anesthetist who performed the anesthesia and the investigators who gathered the data were blinded to patients' group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): PCA ketamine (Ketamine HCl, Pfizer Inc., US) 0.5 mg plus morphine 0.5 mg ml-1 (ratio 1:1) as postoperative analgesia.
  Interventions: Drug: Ketamine-Morphine
- Group B (Active Comparator): PCA morphine (Pfizer Inc., US) 1 mg ml-1 as postoperative analgesia.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ketamine-Morphine — PCA ketamine (Ketamine HCl, Pfizer Inc., US) 0.5 mg plus morphine 0.5 mg ml-1 (ratio 1:1)
  Other Names: Ketamine Hydrochloric, Pfizer Inc., US; Morphine Pfizer Inc., US
  Arms: Group A
Drug: Morphine — PCA morphine (Pfizer Inc., US) 1 mg ml-1
  Other Names: Morphine Pfizer Inc., US
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of PCA ketamine-morphine versus conventional PCA morphine in postoperative patients undergoing elective laparotomy colorectal surgery under general anaesthesia. The specific objectives are:

1. To compare the postoperative analgesic requirement with PCA ketamine-morphine in comparison with PCA morphine.
2. To compare the postoperative pain scores between PCA ketamine-morphine and PCA morphine.
3. To assess patients' overall satisfaction with PCA ketamine-morphine in comparison with PCA morphine.
4. To study the incidence of side effects of PCA ketamine-morphine in comparison with PCA morphine.

Participants will be screened and recruited at the pre-anaesthetic clinic (PAC). Those who consented will be taught to use the PCA machine and the potential side effects of the study drugs. They will be randomly allocated into either Group A or Group B by computer-generated randomization a day before planned surgery.

Researchers will compare Group A and Group B to see post-operative pain scores, patients' overall satisfaction and any incidence of side effects.

DETAILED DESCRIPTION:
INTRODUCTION

Patient-controlled analgesia (PCA) has been an established efficient and safe technique for providing postoperative analgesia [1-3]. It is a delivery system with which patients self-administer predetermined doses of analgesic medication to relieve their pain [1]. A reviewed meta-analysis conducted by McNicol et al (2015) provided evidence that PCA opioids provide superior analgesia in comparison to conventional intravenous opioids analgesia [2]. PCA has been associated with better pain relief and patient satisfaction with less postoperative complications and side effects [1-3].

Despite years of advances in pain management, opioids have been the mainstay for the treatment of postoperative pain particularly in moderate to severe pain [1-3]. A variety of opioids have been used for PCA, namely morphine, fentanyl, pethidine and oxycodone. Of all the opioids, morphine is the most studied drug and remained the drug of choice for PCA including in Malaysian hospitals' settings [1,4]. However, it is also associated with known side effects such as respiratory depression, sedation, nausea and vomiting, pruritus, constipation and urinary retention [2,4]. The concept of multimodal analgesia hence was introduced to reduce opioid-related side effects. Adjuvants such as acetaminophen and non-steroidal anti-inflammatory drugs are commonly used nowadays in combination with opioids as opioid-sparing agents [5, 6].

Ketamine, an N-methyl-D-aspartate (NMDA) antagonist, has undergone a recent resurgence of interest among acute care providers as an adjunct in acute pain management [5-7]. Ketamine at sub-anaesthetic dose (0.2-0.5 mg/kg) produces intense analgesia [5-9]. The analgesic effects of ketamine are primarily due to its activity in the thalamic and limbic systems which are responsible for interpretation of painful signals and modulation of pain [9]. Activation of NMDA receptors located at the dorsal horns, by excitatory neurotransmitters particularly glutamate, induced by peripheral nociceptive stimuli results in hyperexcitability of the dorsal root neurones, which is the pathophysiology of acute pain. It has also been reported that μ receptor activation by opioids leads to a sustained increase in glutamate synaptic effectiveness at the level of NMDA receptors [8]. The combination of ketamine, a non-competitive antagonist at the NMDA receptor with morphine hence will have a synergistic effect and this may allow a reduction in doses of both drugs and potentially reduce the side effects related to both [8-18].

Since its development in 1962, various studies have been conducted to prove the efficacy of ketamine as postoperative analgesia and as an opioid-sparing agent [7]. A review by Laskowski et al. (2010) described IV ketamine improved the quality of pain control, in addition to decreased opioid consumption with particular benefits observed in painful procedures, including upper abdominal, thoracic, and major orthopaedic surgeries [7]. Carstensen et al. (2010) in a qualitative review comparing PCA ketamine-morphine with PCA morphine alone also described the superior efficacy of ketamine-morphine in providing pain control with a significantly higher incidence of opioid-related side effects including sedation, nausea, vomiting, pruritus, urinary retention and desaturation in the morphine group [10]. In comparison to opioids, ketamine's lack of respiratory depressant effects also favours its use as an opioid adjunct in patients with airway and respiratory compromise, such as morbid obesity and post-thoracotomy patients [7,10-13].

The main concern and limitation with regard to ketamine use is its psychomimetic side effects, particularly hallucinations and delirium. However, most studies suggested that the incidence of psychomimetic side effects is minimal with a subanaesthetic dose of ketamine. Both Subramaniam et al. (2004) and Carstensen et al. (2010) found no significance increased in CNS and psychomimetic side effects in patients receiving ketamine as compared to morphine alone [8,11]. While Mathews et al. (2012) reported an incidence of hallucination/vivid dreams requiring the intervention of 2.9%, and an incidence requiring no intervention of 3.3% in a prospective cohort study of 1026 patients receiving PCA ketamine-morphine post-operatively in a variety of surgical settings [12]. The optimum dose for ketamine in combination with morphine is also another issue being addressed in most studies, as various studies used different doses and combinations of ketamine with morphine. A study conducted by Sveticic et al. (2003) analysed 12 different combinations of ketamine and morphine in PCA and their correlation with reduction in pain score and incidence of side effects following spine and hip surgery. The study recommended a combination of morphine with ketamine in a ratio of 1:1 as the best ratio [18].

Despite the potential efficacy with published evidence of PCA ketamine-morphine in postoperative pain management, its use is not well established in most Malaysian hospitals including Hospital Sultanah Aminah Johor Bahru. The use of PCA ketamine however, has been practised in selective postoperative abdominal surgery patients in our Intensive Care Unit (ICU) setting, owing to the fact that ketamine is superior to opioids in reducing the risk of postoperative ileus and nausea and vomiting which may already be exacerbated by the patient's underlying illnesses. The PCA ketamine regime used in our ICU is 1mg/ml bolus with a lock-out period of 5 minutes and background infusion of 1mg/hour, which is, as per our experience, well tolerated in most patients. Therefore, hopefully, the results gained from this study will help us to understand better about PCA ketamine-morphine and its effectiveness in our local population, in the hope that we can provide better care and postoperative pain management for our patients in the future.

METHODS

This prospective double-blind randomized controlled trial was conducted in Hospital Sultanah Aminah Johor Bahru from February to October 2018 after obtaining ethics approval from the local and institutional ethics committee (NMRR-17-1863-37291 & JEP-2018-092). Sixty elective American Society of Anaesthesiologists (ASA) I or II patients scheduled for lower midline laparotomy colorectal surgery aged between 18-70 years old were recruited and informed consent were obtained. All patients who consented were taught the usage of a PCA machine and the potential side effects of ketamine and morphine preoperatively. They were randomly allocated into either Group A or Group B by computer-generated randomization a day before planned surgery.

Group A received PCA ketamine (Ketamine HCl, Pfizer Inc., US) 0.5 mg plus morphine 0.5 mg ml-1 (ratio 1:1) while Group B received PCA morphine (Pfizer Inc., US) 1 mg ml-1 as postoperative analgesia. There was no baseline infusion and the lock-out period was set to 5 minutes. The study drugs were prepared one day before the surgery by the pharmacist who was not involved in the intraoperative and postoperative management of the patients. The drugs were labelled as study drugs with the study number. The patients, nurses who cared for the patients, the anaesthetist who performed the anaesthesia and the investigators who gathered the data were blinded to patients' group allocation.

All patients had standard monitoring of blood pressure, electrocardiogram (ECG), oxygen saturation and end-tidal carbon dioxide (CO2). They were pre-oxygenated with 100% oxygen for 2-3 minutes. The induction of general anaesthesia was standardized to intravenous (IV) fentanyl (Cephalon Inc., US) 2 mcg kg-1, IV propofol (Diprivan, Pfizer Inc., US) 2 mg kg-1 and IV rocuronium (US) 0.6 mg kg-1 and intubation with the appropriate size of the endotracheal tube. Anesthesia was maintained with desflurane (Suprane, Novartis AG, Switzerland) in a mixture of 50% of oxygen and 50% of air, and titrated to achieve a minimum alveolar concentration (MAC) of 1.0. All patients received IV dexamethasone (US) 8 mg after induction and IV morphine 0.1 mg kg-1 as intraoperative analgesia. Boluses of IV fentanyl 25 mcg were given if extra analgesia was required and recorded. IV ondansetron (US) 4 mg was given upon initiation of skin closure. The skin incision site was infiltrated with 0.25% Bupivacaine (US) 10-20 ml during skin closure. The standard dose of IV neostigmine and IV atropine was used to reverse residual neuromuscular blockade at the end of surgery.

At the recovery bay, pain score was assessed using the Numerical Rating Scale (NRS), by which patients scored their pain intensity between number 0 to 10, with 0 being no pain at all and 10 being the worst pain imaginable. If the pain score was > 4 at rest, IV morphine boluses were given and titrated according to the pre-set morphine protocol until the pain score was ≤ 4. PCA machine with the study drug(s) was commenced once the pain score was ≤ 4 at rest.

Patients were assessed 30 minutes after the commencement of PCA, at 6 hourly intervals for the first 24 hours and subsequently at 12 hourly intervals for the next 24 hours post-operatively by the Acute Pain Service (APS) team. They were solely on PCA as post-operative analgesia as the patients were kept nil by mouth for the first 48 hours postoperatively. All patients were assessed for pain score, sedation score, respiratory rate and other side effects of morphine and ketamine including nausea and vomiting, pruritus, dizziness and hallucinations. If the pain score was > 4 at rest during the assessment, 2 ml of PCA drug was given as boluses and titrated every 10 minutes to achieve a pain score ≤ 4.

Cumulative morphine consumption was also recorded. Sedation was assessed using Pasero Opioid-Induced Sedation Scale (POSS) (S - sleep, easy to arouse, 1 - awake and alert, 2 - slightly drowsy, easy to arouse, 3 - frequently drowsy, arousable, drift to sleep during the conversation, 4 - somnolent, minimal or no response to verbal or physical stimulation). Treatment for nausea, vomiting and pruritus was given as deemed appropriate and recorded. At 48 hours post-operation, the patient's overall satisfaction score was assessed using a 1 to 5 Likert scale (1 - very unsatisfied, 2 - unsatisfied, 3 - neutral, 4 - satisfied and 5 - very satisfied). If patients experience hallucinations or delirium, the PCA bolus dose was reduced by 0.2 ml and the symptoms were reassessed after 1 hour. If symptoms persist, the PCA bolus dose was reduced further by 0.2 ml every hour until symptoms disappear and PCA subsequently continued at the reduced dose.

Patients with complicated surgeries in which they became haemodynamically unstable and required post-operative ICU admission, developed anaphylaxis after commencement of study drugs, developed persistent delirium or hallucination after reduction of PCA bolus dose and pain was uncontrollable with the reduced dose or those who refused to continue with the study for any reasons were withdrawn from the study and given other means of analgesia as appropriate by the acute pain service (APS) team.

The sample size was calculated using the Power and Sample Size Calculations program. The α value is set at 0.05 and the power of study at 90%. The sample size is calculated using a t-test. The calculation is derived from the mean pain score and standard deviation as quoted in Javery et al. [12].

Requested output: Sample size

Independent:

Alpha = 0.05; power = 0.9; δ = 1.5; SD 1.67 The case sample size for the t-test = 27 Total sample: 27 x 2 plus 10% drop-out rate = 60 Sample = 30 per study group

All data were analyzed using the SPSS (Statistical Package for The Social Sciences) software. The chi-square test or Fisher exact test was used when appropriate to calculate any significant differences for categorical variables. An Independent t-test or Mann-Whitney U test was used as appropriate to determine any significant differences for continuous variables. The incidence of side effects between the two groups was compared using the Chi-square test. A p-value of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) I or II patients.
2. Patients between 18- 70 years of age.
3. Patients undergoing elective laparotomy colorectal surgery.

Exclusion Criteria:

1. Patients with a known allergy to morphine or ketamine.
2. Patients with uncontrolled hypertension.
3. Patients with a past history of chronic pain on regular analgesics.
4. Patients on psychiatric drugs.
5. Patients with BMI more than 35.
6. Patients with Creatinine Clearance < 30

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
PCA drugs demanded and delivered | 30 minutes after commencement of PCA until 48 hours
  Total PCA drugs demanded and delivered
Pain score | 30 minutes after commencement of PCA until 48 hours
  Pain score at rest and on movement with NRS
  Numerical Rating Scale (NRS) for pain score assessment A numerical pain assessment tool from 0 to 10, where 0 denotes no pain, 5 denotes moderate pain and 10 denotes worst possible pain.
Incidence of side effects | 30 minutes after commencement of PCA until 48 hours
  Opiod related side effects : nausea and vomiting, pruritus, dizziness, respiratory depression and treatment on PRN basis if indicated Ketamine related side effects : delirium, hallucinations, hypertension, tachycardia
Patients' overall satisfaction | At 48 hours post operative
  Assessment of patients' overall satisfaction with a 5-points scales at 48 hours.
  A 5-point scale from 1 to 5, where:
  * very unsatisfied
  * unsatisfied
  * neutral
  * satisfied
  * very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Yong C Liu, MMed (Anaes), Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Momeni M, Crucitti M, De Kock M. Patient-controlled analgesia in the management of postoperative pain. Drugs. 2006;66(18):2321-37. doi: 10.2165/00003495-200666180-00005. PMID 17181375
- [Background] McNicol ED, Ferguson MC, Hudcova J. Patient controlled opioid analgesia versus non-patient controlled opioid analgesia for postoperative pain. Cochrane Database Syst Rev. 2015 Jun 2;2015(6):CD003348. doi: 10.1002/14651858.CD003348.pub3. PMID 26035341
- [Background] Macintyre PE. Safety and efficacy of patient-controlled analgesia. Br J Anaesth. 2001 Jul;87(1):36-46. doi: 10.1093/bja/87.1.36. No abstract available. PMID 11460812
- [Background] Dolin SJ, Cashman JN. Tolerability of acute postoperative pain management: nausea, vomiting, sedation, pruritus, and urinary retention. Evidence from published data. Br J Anaesth. 2005 Nov;95(5):584-91. doi: 10.1093/bja/aei227. Epub 2005 Sep 16. PMID 16169893
- [Background] Argoff CE. Recent management advances in acute postoperative pain. Pain Pract. 2014 Jun;14(5):477-87. doi: 10.1111/papr.12108. Epub 2013 Aug 15. PMID 23945010
- [Background] Vadivelu N, Mitra S, Narayan D. Recent advances in postoperative pain management. Yale J Biol Med. 2010 Mar;83(1):11-25. PMID 20351978
- [Background] Laskowski K, Stirling A, McKay WP, Lim HJ. A systematic review of intravenous ketamine for postoperative analgesia. Can J Anaesth. 2011 Oct;58(10):911-23. doi: 10.1007/s12630-011-9560-0. Epub 2011 Jul 20. PMID 21773855
- [Background] Subramaniam K, Subramaniam B, Steinbrook RA. Ketamine as adjuvant analgesic to opioids: a quantitative and qualitative systematic review. Anesth Analg. 2004 Aug;99(2):482-95, table of contents. doi: 10.1213/01.ANE.0000118109.12855.07. PMID 15271729
- [Background] Stoetling RK, Hiller SK. Pharmacology & Physiology in Anesthetic Practice. 4th edition. Philadelphia: Lippincott Williams & Wilkins. 2006.
- [Background] Carstensen M, Moller AM. Adding ketamine to morphine for intravenous patient-controlled analgesia for acute postoperative pain: a qualitative review of randomized trials. Br J Anaesth. 2010 Apr;104(4):401-6. doi: 10.1093/bja/aeq041. Epub 2010 Mar 5. PMID 20207747
- [Background] Michelet P, Guervilly C, Helaine A, Avaro JP, Blayac D, Gaillat F, Dantin T, Thomas P, Kerbaul F. Adding ketamine to morphine for patient-controlled analgesia after thoracic surgery: influence on morphine consumption, respiratory function, and nocturnal desaturation. Br J Anaesth. 2007 Sep;99(3):396-403. doi: 10.1093/bja/aem168. Epub 2007 Jun 18. PMID 17576969
- [Background] Mathews TJ, Churchhouse AM, Housden T, Dunning J. Does adding ketamine to morphine patient-controlled analgesia safely improve post-thoracotomy pain? Interact Cardiovasc Thorac Surg. 2012 Feb;14(2):194-9. doi: 10.1093/icvts/ivr081. Epub 2011 Nov 28. PMID 22159259
- [Background] Kamal HM. Ketamine as an Adjuvant to Morphine for Patient Controlled Analgesia in Morbidly Obese Patients. Journal of Medical Sciences 2008; 8: 364-370.
- [Background] Javery KB, Ussery TW, Steger HG, Colclough GW. Comparison of morphine and morphine with ketamine for postoperative analgesia. Can J Anaesth. 1996 Mar;43(3):212-5. doi: 10.1007/BF03011736. PMID 8829857
- [Background] Zakine J, Samarcq D, Lorne E, Moubarak M, Montravers P, Beloucif S, Dupont H. Postoperative ketamine administration decreases morphine consumption in major abdominal surgery: a prospective, randomized, double-blind, controlled study. Anesth Analg. 2008 Jun;106(6):1856-61. doi: 10.1213/ane.0b013e3181732776. PMID 18499623
- [Background] Akhavanakbari G, Mohamadian A, Entezariasl M. Evaluation the effects of adding ketamine to morphine in intravenous patient-controlled analgesia after orthopedic surgery. Perspect Clin Res. 2014 Apr;5(2):85-7. doi: 10.4103/2229-3485.128028. PMID 24741486
- [Background] Dahi-Taleghani M, Fazli B, Ghasemi M, Vosoughian M, Dabbagh A. Effect of intravenous patient controlled ketamine analgesiaon postoperative pain in opium abusers. Anesth Pain Med. 2014 Feb 15;4(1):e14129. doi: 10.5812/aapm.14129. eCollection 2014 Feb. PMID 24701419
- [Background] Sveticic G, Gentilini A, Eichenberger U, Luginbuhl M, Curatolo M. Combinations of morphine with ketamine for patient-controlled analgesia: a new optimization method. Anesthesiology. 2003 May;98(5):1195-205. doi: 10.1097/00000542-200305000-00023. PMID 12717142